CLINICAL TRIAL: NCT05165004
Title: Effect of Kangaroo Mother Care Versus Hammock Positioning on Physiological Indices and Behavioral Organization Among Preterm Neonates: A Humanized Nursing Approach
Brief Title: Effect of Kangaroo Mother Care Versus Hammock Positioning
Acronym: Kangaroo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Zohour Ibrahim Mahmoud Rashwan, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2218112020
Record Dates: First submitted 2021-11-25; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Behavior, Child
Keywords: Kangaroo-Mother Care Method; Patient Positioning; Infant Behavior; Physiological; Premature; Neonatal Nursing
MeSH Terms: conditions — Child Behavior; Infant Behavior; Premature Birth | interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kangaroo Mother Care (Experimental): Researchers contacted the mother a day before applying KMC, and advised her to take shower and abstain from using perfumes before attending to the NICU. On days of KMC application, the researchers asked the mother to remove the upper clothes in a private room and put on an open-front gown and mask. The mother was assisted to sit in a comfortable chair with a soft backrest and footrest to prevent fatigue. Then, the preterm neonate was carefully put naked except for the head and diaper area on the mothers' bare chest with flexed arms and legs as in froglike position, and the head was turned sideways. The researchers wrapped and secured the mother's gown and put a blanket on the neonates' back to ensure neonatal thermal insulation. The mother was instructed to support the neonate's bottom with the right hand while supporting the head and neck with the other hand.
  Interventions: Behavioral: Kangaroo Mother Care
- Hammock Positioning (Experimental): Researchers made a hammock by using a rectangular cotton cloth with ropes that passed through the circular openings of the incubator and tied on the upper part of it. After one hour of feeding, the preterm neonate was placed in a supine fetal position in the hammock where the head was supported in a neutral midline position by using rolled towel without neck hyperflexion or hyperextension. Moreover, the spine of the preterm neonate was supported while arms and knees were flexed.
  Interventions: Behavioral: Hammock Positioning
- NICU Routine Care (Active Comparator): The preterm neonates in the control group received the routine care of the NICU, which entails; encircling the neonate in a fetal position using rolled towel inside the incubator.
  Interventions: Behavioral: Routine Care of NICU

INTERVENTIONS:
Behavioral: Kangaroo Mother Care — the preterm neonate was carefully put naked except for the head and diaper area on the mothers' bare chest with flexed arms and legs as in froglike position, and the head was turned sideways. The researchers wrapped and secured the mother's gown and put a blanket on the neonates' back to ensure neonatal thermal insulation
  Arms: Kangaroo Mother Care
Behavioral: Hammock Positioning — After one hour of feeding, the preterm neonate was placed in a supine fetal position in the hammock where the head was supported in a neutral midline position by using rolled towel without neck hyperflexion or hyperextension. Moreover, the spine of the preterm neonate was supported while arms and knees were flexed
  Arms: Hammock Positioning
Behavioral: Routine Care of NICU — ; encircling the neonate in a fetal position using rolled towel inside the incubator.
  Arms: NICU Routine Care

SUMMARY:
Aim

This study aimed to investigate the effect of kangaroo mother care (KMC)versus hammock positioning (HP) on physiological indices and behavioral organization among preterm neonates.

Hypotheses

Preterm neonates who receive KMC exhibit more stable physiological indices and behavioral organization state than those who do not .

Preterm neonates who receive HP exhibit more stable physiological indices and behavioral organization state than those who do not .

Preterm neonates who receive KMC exhibit more stable physiological indices and behavioral organization state than those who receive HP.

DETAILED DESCRIPTION:
A quasi-experimental, pre-posttests, research design was carried out at the Neonatal Intensive Care Unit (NICU) of Specialized University Hospital . A sample of 90 preterm neonates were randomly assigned into three equal groups. The preterm neonates in the control group received the routine care of the NICU, which entails; encircling the neonate in a fetal position using rolled towel inside the incubator.

For the KMC group:

Researchers contacted the mother a day before applying KMC, and advised her to take shower and abstain from using perfumes before attending to the NICU. On days of KMC application, the researchers asked the mother to remove the upper clothes in a private room and put on an open-front gown and mask. The mother was assisted to sit in a comfortable chair with a soft backrest and footrest to prevent fatigue. Then, the preterm neonate was carefully put naked except for the head and diaper area on the mothers' bare chest with flexed arms and legs as in froglike position, and the head was turned sideways. The researchers wrapped and secured the mother's gown and put a blanket on the neonates' back to ensure neonatal thermal insulation. The mother was instructed to support the neonate's bottom with the right hand while supporting the head and neck with the other hand.

For HP group:

Researchers made a hammock by using a rectangular cotton cloth with ropes that passed through the circular openings of the incubator and tied on the upper part of it. After one hour of feeding, the preterm neonate was placed in a supine fetal position in the hammock where the head was supported in a neutral midline position by using rolled towel without neck hyperflexion or hyperextension. Moreover, the spine of the preterm neonate was supported while arms and knees were flexed.

Kangaroo mother care and HP were performed in the morning shift for one hour from 10 am till 11 am on three consecutive days. Behavioral states of preterm neonates were assessed in the three groups four times during the intervention at fixed intervals in order to minimize the measurement errors due to fluctuations in their behavioral states. In case of incidental neonatal distress, the intervention was discontinued. After one hour of applying KMC or HP, the preterm neonates were placed in the incubator as the routine NICU care. Finally, neonates' physiological indices and behavioral states in the three groups were recorded after 15 min from the intervention using tools I&II. Data were collected over 12 months from March 2020 till the end of February 2021.

ELIGIBILITY:
Inclusion Criteria:

* Preterm Neonates
* Hemodynamically stable

Exclusion Criteria:

* Mechanically Ventilated
* Pulmonary Disorders
* Cardiac Disorders,
* Neurological Disorders

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-23 (Actual)

PRIMARY OUTCOMES:
Neonates' Heart Rate (HR) | immediately after the intervention
  The researchers recorded the neonates' heart rate from the ECG monitor
Neonates' Respiratory Rate (RR) | immediately after the intervention
  The researchers recorded the neonates' Respiratory Rate (RR) the ECG monitor
Neonates' Oxygen Saturation (SpO2) | immediately after the intervention
  The researchers recorded the neonates' oxygen saturation (SpO2) using the pulse oximetry
Neonates' Temperature | immediately after the intervention
  The researchers measure the neonates' temperature using electronic thermometer
Neonates' Weight | 3 days After the intervention
  The researchers measure the neonates' weight using digital weighing scale
Anderson Behavioral State Scale | immediately after the intervention
  This scale was adopted from Anderson et al. (1990) to assess the behavioral organization of preterm neonates. Neonates' behavioral state is judged by observing their respiratory regularity, opening or closing of the eyes, limb and trunk activity, and the intensity of crying. Based on the observations, the scale will differentiate 12 behavioral states, including; regular quiet sleep (1), irregular quiet sleep (2), active sleep (3), very active sleep (4), drowsy (5), alert inactivity (6), quite awake (7), active awake (8), very active awake (9), fussing (10), crying (11) and hard crying (12). Scores from 1 to 5 indicate that the neonate is in a sleep state. Scores from 6 to 8 denotes that the neonate is awake and calm. Scores from 9 to 12 indicate that the neonate is in a restless state of or fussiness.

CONTACTS AND LOCATIONS:
Overall Officials: Eman m Taha, professor, Study Chair — Alexandria University
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Farrash RA, Shinkar DM, Ragab DA, Salem RM, Saad WE, Farag AS, Salama DH, Sakr MF. Longer duration of kangaroo care improves neurobehavioral performance and feeding in preterm infants: a randomized controlled trial. Pediatr Res. 2020 Mar;87(4):683-688. doi: 10.1038/s41390-019-0558-6. Epub 2019 Sep 7. PMID 31493775
- [Background] Campbell-Yeo ML, Disher TC, Benoit BL, Johnston CC. Understanding kangaroo care and its benefits to preterm infants. Pediatric Health Med Ther. 2015 Mar 18;6:15-32. doi: 10.2147/PHMT.S51869. eCollection 2015. PMID 29388613
- [Background] Feldman R, Rosenthal Z, Eidelman AI. Maternal-preterm skin-to-skin contact enhances child physiologic organization and cognitive control across the first 10 years of life. Biol Psychiatry. 2014 Jan 1;75(1):56-64. doi: 10.1016/j.biopsych.2013.08.012. Epub 2013 Oct 4. PMID 24094511
- [Background] Jesus VR, Oliveira PMN, Azevedo VMGO. Effects of hammock positioning in behavioral status, vital signs, and pain in preterms: a case series study. Braz J Phys Ther. 2018 Jul-Aug;22(4):304-309. doi: 10.1016/j.bjpt.2018.03.002. Epub 2018 Mar 15. PMID 29598896
- [Background] Korraa AA, El Nagger AA, Mohamed RA, Helmy NM. Impact of kangaroo mother care on cerebral blood flow of preterm infants. Ital J Pediatr. 2014 Nov 13;40:83. doi: 10.1186/s13052-014-0083-5. PMID 25391600
- [Background] Menger JL, Mafaldo LR, Schiwe D, Schaan CW, Heinzmann-Filho JP. EFFECTS OF HAMMOCK POSITIONING ON CLINICAL PARAMETERS IN PRETERM INFANTS ADMITTED TO A NEONATAL INTENSIVE CARE UNIT: A SYSTEMATIC REVIEW. Rev Paul Pediatr. 2020 Nov 30;39:e2019399. doi: 10.1590/1984-0462/2021/39/2019399. eCollection 2020. PMID 33263617